CLINICAL TRIAL: NCT00142220
Title: Comparison Between Two Different Proportions of Omega-3- and Omega-6-Fatty Acids in the Parenteral Nutrition of Critically Ill Patients
Brief Title: The Benefit of Adding Fish Oil to the Nutrition of Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Fresenius AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMEGAVEN
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Sepsis Syndrome
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

INTERVENTIONS:
Drug: Defined percentage of omega-3-fatty acids

SUMMARY:
We study whether an increased proportion of omega-3-fatty acids (contained in fish oil) in the nutrition of critically ill patients reduces systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* indication for parenteral nutrition

Exclusion Criteria:

* hypertriglyceridemia
* coagulation disorder
* decompensated liver cirrhosis or acute liver failure

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160
Dates: Start 2004-01

PRIMARY OUTCOMES:
level of IL-6 in serum
HLA-expression on monocytes

SECONDARY OUTCOMES:
number of nosocomial infections
days on mechanical ventilation
duration of ICU stay
mortality
SOFA score

CONTACTS AND LOCATIONS:
Overall Officials: Sigrun Friesecke, Dr., Principal Investigator — University Medicine Greifswald
Locations (1):
- Internistische ITS, Greifswald, Germany